CLINICAL TRIAL: NCT03039413
Title: Targeting a Genomic Biomarker for PET Imaging and Staging of Urothelial Cancer: A Preliminary Evaluation
Brief Title: Copper Cu-64 TP3805 PET/CT in Imaging Patients With Urothelial Cancer Undergoing Surgery or Biopsy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16G.500; JT 9148 (Other: JeffTrial Number)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Bladder Urothelial Carcinoma; Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Copper Cu 64 TP3805 PET/CT) (Experimental): Patients receive copper Cu 64 TP3805 IV and undergo PET/CT after 60 minutes. Patients then undergo standard of care cystectomy and/or biopsy 1 to 4 weeks later.
  Interventions: Drug: Copper Cu 64 TP3805; Procedure: Positron Emission Tomography; Procedure: Computed Tomography

INTERVENTIONS:
Drug: Copper Cu 64 TP3805 — Given IV
  Other Names: Cu-64-TP3805
Procedure: Positron Emission Tomography — Undergo Cu-64-TP3805 Positron Emission Tomography scan
  Other Names: Medical Imaging; PET; Positron Emission Tomography Scan
Procedure: Computed Tomography — Undergo Cu-64-TP3805 Computed Tomography scan
  Other Names: CAT; Computerized Axial Tomography; CAT scan

SUMMARY:
This pilot clinical trial studies how well copper Cu-64 TP3805 positron emission tomography (PET)/computed tomography (CT) works in imaging patients with urothelial cancer undergoing surgery or biopsy. Radioactive tracers, such as copper Cu-64 TP3805, may bind to tumor cells. PET/CT imaging performed with copper Cu-64 TP3805 may be a better way to detect urothelial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if copper Cu-64 TP3805 (Cu-64-TP3805) shall image urothelial carcinoma (UC) as confirmed by postsurgical or biopsy histology.

SECONDARY OBJECTIVES:

I. To determine blood clearance of Cu-64-TP3805. II. To determine in vivo stability of Cu-64-TP3805.

TERTIARY:

I. To determine if Cu-64-TP3805 is bound to malignant cells and if it is internalized.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Must have diagnosis of urothelial cancer
* Scheduled for extirpative surgery or biopsy of suspected metastatic lesion
* Women of reproductive potential must have a urine pregnancy test day of injection
* Men of reproductive potential must use condoms

Exclusion Criteria:

* Pregnancy or lactation
* Known allergic reactions to components of the study product(s)
* Treatment with another investigational drug or other intervention with 24 hours of injection
* Must not have had an injection of a radioisotope 24 hours prior to exam

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Feasibility of Cu-64-TP3805 to detect UC as determined by post-surgical histology | Up to 4 weeks post-intervention
  For imaging, positive lesions will be deemed those which shall have standard uptake volume of 1.1 or greater. The results shall be correlated with post-surgical histology

SECONDARY OUTCOMES:
Blood clearance defined as the point at which radioactivity decreases to 50% of the initial value | Up to 120 minutes post injection
  The blood clearance time from all subjects shall be averaged with standard error of the mean.
Radioactivity internalization of copper Cu 64 TP3805 as analyzed in centrifuged urine samples | Up to 120 minutes post injection
  Radioactivity associated with supernatant containing cell cytoplasmic component to and cell membrane button shall be counted and their respective percentage shall be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Thakur, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/